CLINICAL TRIAL: NCT01836458
Title: An Open-label Study to Find the Minimum Inhibitory Concentration(MIC) of KAE609 in Adult Male Patients With Acute, Uncomplicated Malaria Due to Plasmodium Falciparum Monoinfection
Brief Title: A Study to Find the Minimum Inhibitory Concentration of KAE609 in Adult Male Patients With P. Falciparum Monoinfection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CKAE609A2201
Record Dates: First submitted 2013-04-17; First posted 2013-04-19 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-09

CONDITIONS: Malaria
Keywords: Malaria, KAE609
MeSH Terms: conditions — Malaria | interventions — NITD 609

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dose 1: 30 mg (Experimental): Single dose of KAE609 30 mg
  Interventions: Drug: KAE609
- Dose 2: 20 mg (Experimental): Single dose of KAE609 20 mg
  Interventions: Drug: KAE609
- Dose 3: 10 mg (Experimental): Single dose of KAE609 10 mg
  Interventions: Drug: KAE609
- Dose 4: 15 mg (Experimental): Single dose of KAE609 15 mg
  Interventions: Drug: KAE609

INTERVENTIONS:
Drug: KAE609 — Patients will receive KAE609 single dose at a different dose level in each cohort.

SUMMARY:
This study aims to determine the Minimum Inhibitory Concentration of KAE609 in adult male patients with acute, uncomplicated malaria due to P.falciparum monoinfection after single dosing with KAE609

DETAILED DESCRIPTION:
There will be a total of approximately 45 patients recruited into this study and six doses of KAE609 and will be investigated.The dose groups will run in sequence. Patient will be given a single dose of KAE609 and be followed up for 42 days.

ELIGIBILITY:
Key Inclusion Criteria:

* Monoinfection with P. falciparum confirmed by microscopy
* Asexual P. falciparum parasitemia count of 5,000 to 50,000/µL
* Axillary temperature ≥37.5 ºC or oral/tympanic/rectal temperature ≥38 ºC; or similar documented temperature during the previous 24 hours
* Body weight between 40 to 90 kg

Key Exclusion Criteria:

* Signs and symptoms of severe malaria according to World Health Organization (WHO) 2010 criteria
* Mixed Plasmodium infection, i.e. infection with more than one species of malaria parasites
* Use of other investigational drugs within 30 days or within 5 half-lives of enrollment, whichever is longer
* History of antimalarial use within 2 months of screening
* Use of any antibiotics with antimalarial activity or other prohibited medication within 14 days of screening
* Long QT syndrome or QTc using Fridericia's formula >430 msec
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases
* Hemoglobin level <10 g/dL
* Liver disease or injury as indicated by elevated liver tests such as SGPT (ALT) or SGOT (AST) >2 times the upper limit of normal
* Renal dysfunction as indicated by serum creatinine >2 times the upper limit of normal in the absence of dehydration; in case of dehydration, serum creatinine should be <2 times the upper limit of normal after oral or parental rehydration
* Known to be immunocompromised (including HIV infection) or are receiving immunosuppressive therapy at the time or enrollment; HIV testing is not required
* Known history of hepatitis B or C; testing is not required
* Febrile condition due to diseases other than malaria (e.g. acute lower respiratory tract infection), known underlying chronic or severe disease (e.g. cardiac, hepatic, renal, gastrointestinal, neurologic, or psychiatric disease), or any condition precluding enrollment into this study according to the investigator
* Severe vomiting defined as >3 times during the previous 24 hours or inability to tolerate oral medication; severe diarrhea defined as ≥3 watery stools during the previous 24 hours
* Severe malnutrition defined by a body mass index (BMI) <18.5 kg/m2 or unintentional loss of weight ≥10% with evidence of suboptimal intake resulting in loss of subcutaneous fat and/or severe muscle wasting
* Active tuberculosis or history of taking anti-tuberculosis medications within 24 months prior to screening

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Ho Chi Minh City, Vietnam

REFERENCES:
- [Derived] Hien TT, White NJ, Thuy-Nhien NT, Hoa NT, Thuan PD, Tarning J, Nosten F, Magnusson B, Jain JP, Hamed K. Estimation of the In Vivo MIC of Cipargamin in Uncomplicated Plasmodium falciparum Malaria. Antimicrob Agents Chemother. 2017 Jan 24;61(2):e01940-16. doi: 10.1128/AAC.01940-16. Print 2017 Feb. PMID 27872070

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dose 1: 30 mg | Dose 2: 20 mg | Dose 3: 10 mg | Dose 4: 15 mg
Started | 7 | 4 | 7 | 7
Completed | 4 | 2 | 2 | 1
Not Completed | 3 | 2 | 5 | 6
Not completed — Unsatisfactory therapeutic effect | 3 | 2 | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose 1: 30 mg | Dose 2: 20 mg | Dose 3: 10 mg | Dose 4: 15 mg | Total
Number analyzed (Participants) | 7 | 4 | 7 | 7 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.7 (11.84) | 32.8 (7.93) | 30.6 (8.24) | 34.7 (8.79) | 32.7 (9.04)
Sex/Gender, Customized [Number; unit: participants]
  MALE | 7 | 4 | 7 | 7 | 25

OUTCOME MEASURES:

1. Primary Outcome: Minimum Inhibitory Concentration (MIC) of KAE609
Description: To observe the exposure-response (PK/PD) relationship for a single dose of KAE609. The key parameter is MIC, defined as the concentration at which the relative rate of change in parasitemia is equal to zero. Approximation of MIC will assist in identifying the optimal dose of KAE609, which will be one component of a future combination antimalarial. MIC could not be determined due to small sample size no data was collected from any participants.
Time Frame: Up to Day 8 after a single dose of KAE609
Population: The primary Outcome Measure (OM) could not be determined due to small sample size no data was collected from any participants.
Arm/Group | Dose 1: 30 mg | Dose 2: 20 mg | Dose 3: 10 mg | Dose 4: 15 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Median Time to Parasite Clearance
Description: Parasite clearance time will be estimated using thick/thin blood films.
Time Frame: pre-dose, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 20, 24, 30, 36, 42, 48, 54, 60, 66, 72 hours post dose of KAE609
Population: Pharmacodynamic Analysis Set includes all enrolled patients
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Dose 1: 30 mg | Dose 2: 20 mg | Dose 3: 10 mg | Dose 4: 15 mg
Number analyzed (Participants) | 7 | 4 | 7 | 7
hours | 24.00 [12.00 to 48.00] | 63.00 [36.02 to 72.00] | 54.00 [36.05 to NA] — Only 4 of 7 patients reached time to parasite clearance; therefore, it was not possible to calculate the upper limit of the 95% confidence interval. | 60.00 [36.00 to 72.00]

3. Secondary Outcome: Median Time to Fever Clearance
Description: Fever is monitored on participants every 4 hours for the first 24 hours, then every 6 hours until negative reading obtained.
Time Frame: Day 1 to Day 5
Population: Pharmacodynamic Analysis Set includes all enrolled patients
Measure: Median (90% Confidence Interval); unit: hours
Arm/Group | Dose 1: 30 mg | Dose 2: 20 mg | Dose 3: 10 mg | Dose 4: 15 mg
Number analyzed (Participants) | 7 | 4 | 7 | 7
hours | 9.83 [0.83 to 11.92] | 12.38 [3.83 to 29.83] | 15.75 [0.75 to 15.83] | 11.83 [4.83 to 35.83]

4. Secondary Outcome: Percentage of Patients PCR-corrected Cure Rate by Day 28, Day 35 & Day 42
Description: PCR-corrected cure rate after a single dose of KAE609 by Day 28, Day 35 & Day 42. PCR-corrected cure rate accounts for failures due to reappearance of parasites that were present in the blood before treatment (i.e. recrudescent infection) but not for failures due to a post-treatment inoculation (i.e. new infection).
Time Frame: Day 28, Day 35 & Day 42
Population: Pharmacodynamic Analysis Set includes all enrolled patients.
Measure: Number; unit: Percentage of Patients
Arm/Group | Dose 1: 30 mg | Dose 2: 20 mg | Dose 3: 10 mg | Dose 4: 15 mg
Number analyzed (Participants) | 7 | 4 | 7 | 7
Percentage of Patients
  Day 28 | 57.1 | 50.0 | 28.6 | 14.3
  Day 35 | 57.1 | 50.0 | 28.6 | 14.3
  Day 42 | 57.1 | 50.0 | 28.6 | 14.3

ADVERSE EVENTS:
Groups:
- Dose 1: 30mg: Single dose of KAE609 30 mg
- Dose 2: 20mg: Single dose of KAE609 20 mg
- Dose 3: 10mg: Single dose of KAE609 10 mg
- Dose 4: 15mg: Single dose of KAE609 15 mg
Arm/Group | Dose 1: 30mg | Dose 2: 20mg | Dose 3: 10mg | Dose 4: 15mg
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/4 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 4/7 | 3/4 | 7/7 | 5/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose 1: 30mg (N=7) | Dose 2: 20mg (N=4) | Dose 3: 10mg (N=7) | Dose 4: 15mg (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abnormal faeces (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 3 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 2 | 3 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.